CLINICAL TRIAL: NCT05422378
Title: A Phase 1 Study to Evaluate the Safety and Tolerability of Subcutaneous Injection of STP705 in Adult Subjects Undergoing Abdominoplasty
Brief Title: A Study to Evaluate Safety, Tolerability of Subcutaneous Injection in Adult Subjects Undergoing Abdominoplasty
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sirnaomics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SRN-705-010
Record Dates: First submitted 2022-06-08; First posted 2022-06-16 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Abdominal Obesity
MeSH Terms: conditions — Obesity, Abdominal | interventions — Injections

STUDY DESIGN:
Intervention Model Description: Dose-ranging, double-blind, vehicle-controlled
Who Masked: Participant, Investigator
Masking Description: double-blind (investigator & subjects)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (7):
- STP705, 120ug/mL, 0.5 cc (Experimental): Volume of Injection 0.5cc
  Interventions: Drug: STP705
- STP705, 120ug/mL, 1.0 cc (Experimental): Volume of Injection 1.0cc
  Interventions: Drug: STP705
- STP705, 240 ug/mL, 0.5 cc (Experimental): Volume of Injection 0.5cc
  Interventions: Drug: STP705
- STP705, 240ug/mL, 1.0 cc (Experimental): Volume of Injection 1.0cc
  Interventions: Drug: STP705
- STP705, 320ug/mL, 0.5 cc (Experimental): Volume of Injection 0.5cc
  Interventions: Drug: STP705
- STP705, 320ug/mL, 1.0 cc (Experimental): Volume of Injection 1.0cc
  Interventions: Drug: STP705
- Vehicle (Placebo Comparator): 1.0cc placebo
  Interventions: Drug: STP705

INTERVENTIONS:
Drug: STP705 — STP705 composed of 2 siRNA targeting TGF-B1and COX-2 individually.
  Other Names: STP705 Powder for Injection

SUMMARY:
Dose-ranging, randomized, double-blind, vehicle-controlled study

DETAILED DESCRIPTION:
Subject will receive a single injection for each treatment which all 3 test article concentrations and both injection volumes and the vehicle for a total of 7 treatments.

Subjects will receive test articles in 3 visits.

ELIGIBILITY:
Inclusion Criteria:

To enter the study, a subject must meet the following criteria:

1. Subject is a male or non-pregnant female 18-65 years of age.
2. Subject has provided written informed consent.
3. Females must be post-menopausal , surgically sterile , or use an effective method of birth control. , Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 3/Baseline.
4. Subject has agreed to undergo an abdominoplasty procedure, participate in this study, has minimally acceptable adipose tissue in the target areas per protocol, and meets all pre-operative requirements, in the opinion of the investigator and surgeon.

Exclusion Criteria:

A subject is ineligible to enter the study if he/she meets one or more of the following criteria:

1. Subject is pregnant, lactating, or is planning to become pregnant during the study.
2. Subject has a significant active systemic or localized abdominal infection.
3. Subject has a body mass index (BMI) ≥40.
4. Subject has any medical condition that affects clotting and/or platelet function (e.g., thromboembolic disease, clotting factor deficiencies such as hemophilia).
5. Subject is taking any medications that affect clotting and/or platelet function. This includes, but is not limited to, heparin (including low molecular weight heparin), Coumadin, and factor Xa agents such as apixaban (Eliquis), etc. The use of such medications is precluded up to 7 days prior to Visit 3/Baseline and during the study period.
6. Subject is immunocompromised, in the opinion of the investigator, based on their medical condition (e.g., HIV positive, malignancy), medication use, or other factors.
7. Subject has any clinically significant medical abnormality or chronic disease of the cardiovascular, gastrointestinal, respiratory (e.g., chronic obstructive pulmonary disease), hepatic, or renal systems. This includes conditions (e.g., gastrointestinal surgery) that may interfere with metabolism or excretion.
8. Subject has local skin condition(s) (e.g., rash, scarring, and tattoos) or inadequate injection sites in the region designated for abdominoplasty excision which are inappropriate for participation in the study, in the opinion of the investigator.
9. Subject is currently enrolled in an investigational drug, biologic, or device study.
10. Subject has used an investigational drug, investigational biologic, or investigational device treatment within 30 days prior to first injection of the test article.
11. Subject has a history of sensitivity to any of the ingredients in the test articles (see Section 6.1).
12. Subject is known to be noncompliant or is unlikely to comply with the requirements of the study protocol (e.g., due to alcoholism, drug dependency, mental incapacity) in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-06-27 (Actual)

PRIMARY OUTCOMES:
Number of subjects with presence and severity of the following Local Skin Reactions (LSR): erythema, edema, bruising. | 24 weeks
  LSR scale will be used by investigator to assess injection site using a 4-point ordinal scale (0=complete absence, 1=mild, limited involvement, 2= moderate involvement, and 3= severe, extreme involvement)
Number of subjects with presence and severity of the following Local Skin Reactions (LSR): pain and stinging/burning. | 24 weeks
  LSR scale will be used by subjects to assess injection site using a 4-point ordinal scale (0=complete absence, 1=mild, 2= moderate, and 3= severe)
Incidence (severity and causality) of any AEs | 24 weeks
  AE's will be classified using CTCAE v.5.0

CONTACTS AND LOCATIONS:
Overall Officials: Mark Nestor, MD, Principal Investigator — Center for Clinical and Cosmetic Research
Locations (1):
- Center for Clinical and Cosmetic Research, Aventura, Florida, United States

REFERENCES:
- [Derived] Nestor MS, Hetzel J, Awad N, Bhupalam V, Lu P, Molyneaux M. A Novel Injectable Polypeptide Nanoparticle Encapsulated siRNA Targeting TGF-beta1 and COX-2 for Localized Fat Reduction II: Phase I Clinical Trial. J Cosmet Dermatol. 2025 Feb;24(2):e16722. doi: 10.1111/jocd.16722. Epub 2024 Dec 18. PMID 39692702